CLINICAL TRIAL: NCT05676749
Title: C-TIL051 in Anti-PD1 Resistant Metastatic Non-Small Cell Lung Cancer
Brief Title: C-TIL051 in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: AbelZeta Inc. (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-2005
Record Dates: First submitted 2022-12-07; First posted 2023-01-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; NKTR-255

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- C-TIL051 (Experimental): C-TIL051 plus IL-15 (NKTR-255) and Pembrolizumab
  Interventions: Biological: C-TIL051

INTERVENTIONS:
Biological: C-TIL051 — C-TIL051 given in combination with IL-15 (NKTR-255) and pembrolizumab
  Other Names: Pembrolizumab; NKTR-255

SUMMARY:
The goal of this Phase 1 clinical study is test tumor infiltrating lymphocytes (known as C-TIL051) with NKTR-255 and anti-PD1 therapy for subjects with refractory non-small cell lung cancer.

The purpose of this study is to:

1. Test the safety and ability for subjects to tolerate the TIL therapy
2. Measure to see how the NSCLC responds to the TIL therapy

Participants will be asked to:

* Provide a tumor sample prior to the start of any treatment which will be used to make the C-TIL051.
* Receive standard of care treatment until their lung cancer no longer responds
* When necessary, the C-TIL051 will be manufactured by the sponsor and sent back to the site
* Subject will then receive chemotherapy (called lymphodepletion) for 3 days followed by 2 days of rest
* C-TIL051 will then be infused on day 0 followed by NKTR-255 (IL-15) about 12 to 24 hours later
* Pembrolizumab will be administered every 3 weeks for up to 2 years

NKTR-255 is a novel polymer-conjugated human IL-15 receptor agonist molecule designed to increase the proliferation and survival of memory CD8+ T cells and enhance the formation of long-term immunological memory which may lead to sustained anti-cancer immune response. The combination of NKTR 255 and TIL's could improve proliferation and persistence of cellular therapies leading to enhanced anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give written informed consent
* Histologically and cytologically confirmed diagnosis of stage IV or recurrent non-small cell lung cancer (NSCLC) with adenocarcinoma or squamous histology
* Planned for treatment with an anti-PD1 agent
* Tumor accessible by surgery, previously not irradiated and ≥ 1.5 cm in diameter
* Measurable disease after resection of tumor by RECIST 1.1
* ECOG ≤ 1
* Expected survival > 6 months
* Adequate organ and marrow function
* ECHO, MUGA or cardiac stress test within past 6 months showing LVEF >50% and without evidence of reversible ischemia
* Pulmonary function tests within past 6 months showing DLCO >50% of predicted

Exclusion Criteria:

* Previous treatment with PD1/PDL1 inhibitor for metastatic disease, Immune checkpoint blockade (ICB) given as part of definitive therapy for stage Ib-III disease with surgery or after chemo/radiation is acceptable if last dose of ICB is at least 6 months prior to enrollment in this study.
* Known driver mutations such as EGFR, ALK, ROS1, RET, METex14, and NTRK alterations.
* Current or prior use of any immunosuppressive medications within 14 days before tumor harvest
* Known active CNS metastases which are symptomatic
* History of leptomeningeal metastases
* Uncontrolled intercurrent illness
* Known history of HIV+ or AIDS, hepatitis C, acute or chronic active hepatitis B or other serious chronic infection
* Live vaccine within 30 days of tumor harvest
* History of allogeneic organ transplant
* History of primary immunodeficiency
* Hypersensitivity to anti-PD1 agent, cyclophosphamide, fludarabine, interleukin-2, gentamicin, or any excipient
* Any condition that may interfere with evaluation of study treatment, safety or study results
* Active infection that requires IV antibiotics within 7 days of tumor harvest
* Unresolved greater than grade 1 toxicity (CTCAE v5.0) from previous therapy
* History of interstitial pneumonitis of autoimmune etiology that is symptomatic or requires treatment
* Pulmonary disease history requiring escalating amounts of oxygen > 2L
* Known autoimmune conditions requiring systemic immune suppression therapy other than low dose prednisone or equivalent.
* Other malignancy, other than cutaneous localized) that required active treatment in the last 2 years.
* Women who are pregnant or lactating
* Women of childbearing potential or fertile men who are unwilling to use effective contraception during study and 6 months after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Calculate the Incidence of Adverse Events or Dose Limiting Toxicities | up to 24 months
  Record the incidence and severity of all adverse events or dose limiting toxicities that occur according to CTCAE criteria V5.0

SECONDARY OUTCOMES:
Calculate Objective Response Rate (ORR) of all Subjects | up to 36 months
  Measure by radiographical imaging (CT/MRI scan) the objective response rate using RECIST 1.1
Calculate Duration of Response (DOR) of All Subjects | up to 36 months
  Measure by radiographical imaging (CT/MRI scan) the length of response in time.
Calculate Progression Free Survival (PFS) for All Subjects | up to 36 months
  Measure by radiographical imaging (CT/MRI scan) the length of time to progression of disease.
Determine Overall Survival (OS) of All Subjects | up to 36 months
  Measure by physical exam and contact reports the overall survival for all subjects following C-TIL051 treatment.

OTHER OUTCOMES:
Collect Blood Samples to Measure the T-cells Before and After C-TIL051 Therapy | up to 24 months
  Collect blood samples to review information about the t-cells present prior to lymphodepleting chemotherapy and after C-TIL051 therapy.
Collect Blood Samples to Measure Cytokines prior to and after C-TIL051 Therapy. | up to 24 months
  Collect blood samples and analyze for presence of cytokines at specified intervals before and after treatment with C-TIL051.
Collect Blood and Tumor Samples to Measure Circulating DNA | up to 24 months
  Collect blood and tumor samples and analyze for circulating DNA.
Collect Blood Samples to Measure Blood RNA | up to 24 months
  Collect blood samples and analyze for RNA sequencing
Perform Radiographic Imaging to Review Antitumor Activity Following Treatment | up to 24 months
  Measure by radiographical imaging (CT/MRI scan) and assess response by immune-related response criteria (irRC).
Collect and Analyze Tumor Samples for MicroOrganoSphereTM (MOS) Technology | up to 36 months
  Collect tumor sample and review outcome measures by MicroOrganoSphereTM (MOS) Technology.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ochsner MD Anderson Cancer Center, New Orleans, Louisiana
  - Duke Center for Cancer Immunotherapy, Raleigh, North Carolina
  - Allegheny Health Network-West Penn Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No